CLINICAL TRIAL: NCT04867499
Title: Retrospective Population-based Study on Epidemiology of Acute Mesenteric Ischemia in Estonia
Brief Title: Epidemiology of Acute Mesenteric Ischemia
Status: Completed | Type: Observational
Sponsor: Tartu University Hospital (Other)
Responsible Party: Principal Investigator, Karri Kase, Medical Doctor, Tartu University Hospital
Other Study IDs: 21021
Record Dates: First submitted 2021-04-20; First posted 2021-04-30 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Acute Mesenteric Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — Descriptive study. No intervention.

SUMMARY:
Retrospective population-based study on epidemiology of acute mesenteric ischemia in Estonia Study objective is to describe epidemiologic features in adult patients with acute mesenteric ischemia during years 2016-2020. Patients from all hospitals in Estonia are included.

ELIGIBILITY:
Inclusion Criteria:

All at least 18-year-old patients with acute mesenteric ischemia during years 2016-2020.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All at least 18-year-old patients with acute mesenteric ischemia during years 2016-2020 in Estonia.
Sampling Method: Non-Probability Sample
Enrollment: 577 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Incidence | 2016-2020
  To identify the incidence of AMI in adult hospitalized patients in Estonia during 2016-2020

CONTACTS AND LOCATIONS:
Locations (1):
- Tartu University Hospital, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kase K, Reintam Blaser A, Tamme K, Mandul M, Forbes A, Talving P, Murruste M. Epidemiology of Acute Mesenteric Ischemia: A Population-Based Investigation. World J Surg. 2023 Jan;47(1):173-181. doi: 10.1007/s00268-022-06805-5. Epub 2022 Oct 19. PMID 36261602

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT04867499/Prot_SAP_000.pdf